CLINICAL TRIAL: NCT01735279
Title: "Studying the Effects of Administration of Polyunsaturated Fatty Acids (PUFAS) of Omega-3 Series in Nicotine Dependence"
Brief Title: Studying the Effects of Administration of Polyunsaturated Fatty Acids (PUFAS) of Omega-3 Series in Nicotine Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Fernandes Galduroz MD, Md PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tobacco&Omega
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Dependence; Nicotine Dependence
Keywords: tobacco dependence; tobacco treatment; omega 3 series; polyunsaturated fatty acids
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Docosahexaenoic Acids; Fish Oils; Fatty Acids, Omega-3; Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo group will receive 3g per day of mineral oil during 90 days treatment
  Interventions: Drug: Placebo
- Omega3 (Experimental): The omega 3 group will receive 3g per day of fish oil during 90 days treatment
  Interventions: Drug: Omega 3

INTERVENTIONS:
Drug: Omega 3 — Each fish oil capsule contained 210.99 mg of EPA and 129.84 mg of DHA.
  Other Names: fish oil; omega 3 fatty acid
  Arms: Omega3
Drug: Placebo — mineral oil + food dye #2 (simulating the colour of essential fatty acids); 1000 mg of mineral oil per capsule
  Other Names: mineral oil
  Arms: Placebo

SUMMARY:
Nicotine dependence may prolong the exposure to toxic substances that cause various diseases. The Central Nervous System (CNS) is consisted by a large amount of Polyunsaturated Fatty Acids (PUFAS) from omega-3 serie. Omega-3 takes part in several actions, including the modulation of dopaminergic neurotransmission. In its deficiency is detected a hypofunctioning of the mesolimbic and mesocortical pathway, related to the reward system, involved on the context of nicotine dependence. Treatment using dietary supplementation with omega-3 shows improvements in several diseases, including mood disorders such as anxiety and depression. The investigators hypothesis is that supplementation with these fatty acids can restore the levels of omega-3 and could decrease nicotine dependence. The investigators objective is to investigate a possible association between increased serum levels of omega-3 and the reduction in nicotine dependence.

DETAILED DESCRIPTION:
Introduction: A cigarette has more than 6,000 toxic substances that can cause various diseases. Nicotine dependence may prolong the exposure to these toxic substances. The Central Nervous System (CNS) is consisted by a large amount of Polyunsaturated Fatty Acids (PUFAS) from omega-3 serie. Omega-3 takes part in several actions, including the modulation of dopaminergic neurotransmission. In its deficiency is detected a hypofunctioning of the mesolimbic and mesocortical pathway, related to the reward system, involved on the context of nicotine dependence. Treatment using dietary supplementation with omega-3 shows improvements in several diseases, including mood disorders such as anxiety and depression. The investigators hypothesis is that supplementation with these fatty acids can restore the levels of omega-3 and could decrease nicotine dependence. Objective: Investigate a possible association between increased serum levels of omega-3 and the reduction in nicotine dependence. Material and Methods: In the clinical study, placebo controlled, double-blind, parallel, randomized, will be administered to 60 volunteers: placebo or fish oil for 90 days. Psychometric assessments will be carried out, measurements of serum levels of PUFAS, levels of carbon monoxide (CO) and cotinine in plasma will be done for monitoring the clinical course. Data Analysis: Repeated measures (ANOVA) for the dependent variables (dependency, anxiety, depression, motivation, compulsion, dosage of PUFAS, exhaled CO and cotinine) and independent (groups and time) to check for significant differences. If so, a second ANOVA with covariates will be conducted. Significance is p <0.05 in all analyzes.

ELIGIBILITY:
Inclusion Criteria:

* healthy smokers; age between 20 and 60 years; score in Fagerström Test for Nicotine Dependence (FTND) up to 5 points (FTND > 5); high motivation to stop smoking (accessed by Richmond Test)

Exclusion Criteria:

* psychiatric disorders; taking psychoactive medications; history of alcohol and/or other drugs abuse or dependence;

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos F. Galduróz, Md PhD, Principal Investigator — Universidade Federal de São Paulo (UNIFESP)
Locations (1):
- Unidade de Dependência de Drogas (UDED), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available. The data obtained was analysed and published

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected in São Paulo/Brazil between January 2013 and August 2013. All participants signed an informed consent prior to the beginning of the study. The participants did not receive any kind of compensation for participation in the study.
Pre-assignment Details: No participants were excluded.
Groups:
- Placebo: placebo capsules 1,000 mg - mineral oil + food dye #2 (simulating the colour of essential fatty acids), taken in 3 daily doses.
- Omega3: omega 3 capsules 1,000 mg fish oil taken as 3 daily doses. Each fish oil capsule contained 210.99 mg of EPA and 129.84 mg of DHA
Period: Overall Study
Arm/Group | Placebo | Omega3
Started | 29 | 29
Completed | 18 | 21
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo capsules 1,000 mg - mineral oil + food dye #2 (simulating the colour of essential fatty acids), taken in 3 daily doses, for 90 days.
- Omega3: omega 3 capsules 1,000 mg fish oil taken as 3 daily doses, for 90 days. Each fish oil capsule contained 210.99 mg of EPA and 129.84 mg of DHA
- Total: Total of all reporting groups
Arm/Group | Placebo | Omega3 | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.5) | 46.2 (11.1) | 47 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 14 | 16 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.7) | 24.7 (3.9) | 24.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Fageström Test for Nicotine Dependence Score at Baseline and After 90 Days of the Treatment
Description: The Fageström Test for Nicotine Dependence is a widely used test to measure the nicotine dependence. This test was chosen to evaluate the possible changes on the nicotine dependence during the clinical trial.
  The range for the scale is:
  very low (dependence) 0-2 low (dependence) 3-4 moderate (dependence) 5 high (dependence) 6-7 very high (dependence) 8-10
  So, lower levels (low scores on the scale) of the FTND measure indicates lower nicotine dependence, and higher levels (high scores on the scales) of the FTND measure indicates higher nicotine dependence.
Time Frame: Baseline (prior to the beginning) and after 90 days of the treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Omega3
Number analyzed (Participants) | 29 | 29
units on a scale
  pre | 6.53 (2.01) | 6.56 (1.52)
  post | 5.96 (1.85) | 5.22 (2.15)

2. Secondary Outcome: Concentration of Docosahexaenoic Acid (DHA) at Baseline and After 90 Days of Treatment
Description: The polyunsaturated fatty acid Docosahexaenoic acid (DHA) is one of the main fatty acids omega-3 series. The dosage of these analyte was achieved by means of Liquid Chromatography - Mass Spectrometry Mass Spectrometry - LS-MS-MS.
Time Frame: At baseline (prior to the beginning of the treatment) and after 90 days of treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Omega3
Number analyzed (Participants) | 29 | 29
ng/ml
  Pre | 747.71 (794.00) | 645.38 (757.49)
  Post | 663.93 (767.41) | 1,004.94 (1,484.63)

3. Secondary Outcome: Concentration of Eicosapentaenoic Acid (EPA)
Description: The polyunsaturated fatty acid Eicosapentaenoic acid (EPA) is one of the main fatty acids omega-3 series. The dosage of these analyte was achieved by means of Liquid Chromatography - Mass Spectrometry Mass Spectrometry - LS-MS-MS.
Time Frame: At baseline (prior to the beginning of the treatment) and after 90 days of treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Omega3
Number analyzed (Participants) | 29 | 29
ng/ml
  Pre | 77.00 (67.72) | 86.76 (111.79)
  Post | 77.39 (73.22) | 174.87 (285.37)

4. Post Hoc Outcome: Concentration of Serum Cotinine at Baseline and After 90 Days of Treatment
Description: Cotinine is the major metabolite of nicotine, making it its primary metabolite. Cotinine dosage is considered one of the best parameters to distinguish smokers from non-smokers as well as for the nicotine graduation consumption. The traditional cut off value used to distinguish between smokers and non-smokers is 15 ng/mL for dosages from plasma sample
Time Frame: At baseline (prior to the beginning of the treatment) and after 90 days of treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Omega3
Number analyzed (Participants) | 29 | 29
ng/ml
  Pre | 101.20 (65.10) | 129.38 (85.15)
  Post | 97.79 (63.26) | 98.54 (61.94)
Statistical Analysis 1: Comparison: Placebo vs Omega3; Test type: Other — Test t Student; p < 0.05, ANOVA; Mean Difference (Final Values) = 0.05
Statistical Analysis 2: Comparison: Omega3; Test type: Superiority; p < 0.01, ANOVA; Mean Difference (Final Values) = 30.84
Statistical Analysis 3: Comparison: Omega3; Test type: Superiority; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = 0.002
Statistical Analysis 4: Comparison: Placebo; Test type: Superiority; p < 0.01, t-test, 1 sided; Mean Difference (Final Values) = 4.4

ADVERSE EVENTS:
Time Frame: The adverse event were collected monthly (after 30, 60 and 90 days of the treatment) during the 90 days (treatment time)
Description: No adverse event were reported by the participants
Groups:
- Placebo Group n= 29: placebo capsules 1,000 mg - mineral oil + food dye #2 (simulating the colour of essential fatty acids), taken in 3 daily doses, for 90 days.
- Omega3 Group n= 29: omega 3 capsules 1,000 mg fish oil taken as 3 daily doses, for 90 days. Each fish oil capsule contained 210.99 mg of EPA and 129.84 mg of DHA
Arm/Group | Placebo Group n= 29 | Omega3 Group n= 29
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No